CLINICAL TRIAL: NCT05780580
Title: Characteristics of Health Insurance Beneficiaries With a Triptan Prescription in the Grand Est Region, France, in 2018-2019 - PASENREGE Study
Brief Title: Prescription of Triptans in the Grand Est Region, France
Acronym: PASENREGE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-02Obs-CHRMT
Record Dates: First submitted 2023-03-10; First posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with a prescription for triptan reimbursed by health insurance
- patients without a prescription for triptan reimbursed by health insurance

SUMMARY:
The high frequency of migraine contrasts with the disparity of its management. The FRAMIG 3 study, carried out in France on the basis of the definition criteria of migraine of the IHS 2004 classification, identified, on the basis of a questionnaire of a representative sample of the general population of 10532 people, 11.2% of the people meeting the criteria of defined migraine and 10.1% of the criteria of probable migraine. Only 40.2% knew they had migraine. 50% used self-medication. Although available since the late 1990s as an effective and specific treatment for migraine attacks, 7.5% of migraineurs in the FRAMIG 3 study used a triptan. In 2003-4, 1.5% of the 1,793,000 inhabitants of Alsace had received at least one prescription for triptans over a one-year period. 1.9% of them were considered overconsumers (greater than or equal to 144 doses/year). More than 10 years later, another population-based study, using data from the French national health agency, identified 1.8% of insured persons receiving a triptan. Several migraine prophylactic treatments have been shown to be effective in patients with frequent or severe migraine attacks, or who do not respond to crisis treatment, or who claim poor quality of life due to migraine, but only 50% of candidates for such prophylactic treatment were receiving it. Only 1.5% of migraine patients in the FRAMIG 3 study were taking prophylaxis. Quality of life was impaired in 57% of migraineurs in the USA and in 28% of French migraineurs. In Ali's study (Ali 2017), 6.9% of migraineurs had used a neurologist. A Brazilian study shows that the average delay of patients accessing a tertiary center was 17 years. As promising new prophylactic treatments become available, we wanted to study a population of migraineurs identified on the basis of a triptan prescription, in order to try to better identify the characteristics of this population, particularly in terms of analgesic consumption and use of specialized care.

The objective of this study was to describe the quantity of triptans dispensed to residents of the Grand Est region aged 12 years and older, between June 1, 2018, and June 1, 2019, based on health insurance data. The secondary objectives were to compare the characteristics of insured persons who had at least one triptan dispensing with those of other insured persons, and to compare the characteristics of insured persons by quantity of triptans dispensed.

ELIGIBILITY:
Inclusion Criteria:

* beneficiary of the general health insurance scheme between june 2018 and june 2019
* at least 12 years old
* resident in the Grand Est region

Exclusion Criteria:

* none

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with migraine
Sampling Method: Non-Probability Sample
Enrollment: 4275652 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
prescription for triptan | 1 year
  Number of insureds with at least one reimbursement for a triptan prescription between June 2018 and June 2019

SECONDARY OUTCOMES:
quantity of triptan consumption | 1 year
  number of boxes of triptans dispensed per insured person, weighted by the number of doses contained per box

CONTACTS AND LOCATIONS:
Overall Officials: Xavier DUCROCQ, MD,, Principal Investigator — CHR Metz Thionville Hopital de Mercy
Locations (1):
- CHR Metz-Thionville/Hopital de Mercy, Metz, France

IPD SHARING:
Plan to Share IPD: No